CLINICAL TRIAL: NCT06142578
Title: Safety and Effectiveness Clinical Evaluation of the Range of Injectable Medical Devices Fillgel in Facial Aesthetic Treatment
Brief Title: Safety and Effectiveness Clinical Evaluation of Injectable Medical Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kylane Laboratoires (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22E0978
Record Dates: First submitted 2023-11-02; First posted 2023-11-21 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Aesthetic Dermatology
Keywords: Aesthetic; dermatology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): FILLGEL 0
  Interventions: Device: Dermal Filler Device
- Group 2 (Experimental): FILLGEL 1
  Interventions: Device: Dermal Filler Device
- Group 3 (Experimental): FILLGEL 2
  Interventions: Device: Dermal Filler Device
- Group 4 (Experimental): FILLGEL 3
  Interventions: Device: Dermal Filler Device

INTERVENTIONS:
Device: Dermal Filler Device — Injection of device by investigators according to the Instruction For Use (IFU)

SUMMARY:
The study aims to confirm the safety and effectiveness of FILLGEL devices

DETAILED DESCRIPTION:
The primary objective is to evaluate the effectiveness of the FILLGEL range used on different treated zones one month (M1) after treatment using clinical evaluation of the global aesthetic improvement (GAIS) rated by the independent investigator. The secondary objectives of the study are to collect data for the

FILLGEL range on:

* the effectiveness of the range used on different treated zones six months (M6) and twelve months (M12) .
* the safety using clinical evaluation of the Injection Site Reactions (ISR) rated by the subject and the investigator.
* subject's satisfaction and subject's opinion on aesthetic improvement on the different treated zones.
* the injector's satisfaction on the injection quality using subjective evaluation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Subject.
2. Sex: male or female.
3. Age: between 18 and 65 years.
4. Subject seeking an improvement of her/his face aspect with Hyaluronic Acid (HA) filler.

   * For group 1: Subject with moderate to severe peri-oral lines (score 3 to 5 on Bazin Upper lip scale) ;
   * For group 2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with thin lips (score

     1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume;
   * For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale);
   * For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement.
5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study.
6. Subject having given their free, express, and informed consent.
7. Subject psychologically able to understand the information related to the study, and to give their written informed consent.
8. Subject registered with a social security scheme.
9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study

Exclusion Criteria:

In terms of population

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject suspected to be non-compliant according to the investigator's judgment.
5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.
6. Subject enrolled in another study or whose non-enrollment period is not over.
7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up…). In terms of associated pathology
8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.
9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria …) in the 6 months before screening visit.
11. Subject with a history of streptococcal disease or an active streptococcus infection.
12. Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kylane Laboratoires, Plan-les-Ouates, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 17 | 17 | 17 | 17
Completed | 17 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 17 | 17 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 57.7 [47 to 65] | 46.7 [20 to 64] | 56.1 [38 to 64] | 54.1 [25 to 64] | 53.6 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 15 | 17 | 64
  Male | 0 | 2 | 2 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 17 | 17 | 17 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Performance
Description: Primary endpoint was the proportion of subjects having an improvement of the zone treated with the overall FILLGEL range of devices, in all the indications, as assessed by the independent investigator, one month after treatment, using the Global Aesthetic Improvement Scale (GAIS) (subjects with a GAIS "improved", "much improved" or "very much improved"). This proportion of responders was compared to a theoretical proportion of 50%.
Time Frame: 1 month
Population: This results is not reported per arm. It is the very purpose of the primary endpoint, to assess the performance of the overall FILLGEL range, independantly of the Arms/groups. The results were not expressed by arms/groups separately, but for the overall FILLGEL range only, as explained in the description: Primary endpoint was the proportion of subjects having an improvement of the zone treated with the overall FILLGEL range of devices, in all the indications...
Measure: Number; unit: percentage of participants
Groups:
- All Groups: FILLGEL 0,1,2,3
Arm/Group | All Groups
Number analyzed (Participants) | 68
percentage of participants | 97.6

2. Secondary Outcome: Performance - GAIS Investigator
Description: Proportion of responders (subjects with a GAIS "improved", "much improved" and "very much improved") for the whole FILLGEL range and by device/indication, with the statistical comparison to the theoretical proportion of 50%.
Time Frame: 6 months, 12 months
Measure: Number; unit: percentage of participants
Arm/Group | All Groups | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 68 | 17 | 17 | 17 | 17
percentage of participants
  At 6 months | 94 | 82.4 | 95.6 | 100 | 96.4
  At 12 months | 88 | 76.5 | 95.6 | 94.1 | 86.8

3. Secondary Outcome: Patients Safety
Description: Proportion of subjects presenting at least one Injection Site Reaction (ISR) evaluated by the investigator, by visit and by indication.
Time Frame: Immediatly after injection (D0), 1 month, 6 months, 12 months
Measure: Number; unit: percentage of at least 1 sign of ISR
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 17 | 17 | 17 | 17
percentage of at least 1 sign of ISR
  Immediatly after injection (D0) | 88 | 100 | 47 | 47
  1 month | 24 | 13 | 6 | 6
  6 months | 0 | 13 | 0 | 0
  12 months | 6 | 0 | 0 | 0

4. Secondary Outcome: Subject Satisfaction - GAIS Subject
Description: Proportion of responders (subjects with a GAIS="improved", "much improved" and "very much improved") for the whole FILLGEL range and by device/indication, with the statistical comparison to the theoretical proportion of 50%.
Time Frame: 1, 6, 12 months
Measure: Number; unit: percentage of participants
Arm/Group | All Groups | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 68 | 17 | 17 | 17 | 17
percentage of participants
  At 1 month | 90.4 | 94.1 | 100 | 100 | 75.3
  At 6 months | 81.9 | 64.7 | 92.9 | 88.2 | 81.2
  At 12 months | 79.5 | 76.4 | 92.9 | 88.1 | 63.3

5. Secondary Outcome: Injector Satisfaction
Description: Distribution of each item of the questionnaire answered by the injectors (injector's satisfaction on the injection quality using subjective evaluation questionnaire).
  The scale is "Very dissatisfied", "Dissatisfied", "Neither satisfied nor dissatisfied", "Satisfied" or "Very satisfied" The percentage of satisfied injectors includes participants that reported being "satisfied" and "very satisfied"
Time Frame: After injection
Measure: Number; unit: percentage of satisfied injectors
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 17 | 17 | 17 | 17
percentage of satisfied injectors
  Easiness of injection | 100 | 100 | 100 | 100
  Easiness of product positionning | 100 | 100 | 100 | 100
  Immediate results | 100 | 100 | 100 | 100
  Result after massage | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Device Under Investigation (Total of Groups): All the groups Group 1: FILLGEL 0 Group 2: FILLGEL 1 Group 3: FILLGEL 2 Group 4: FILLGEL 3
Arm/Group | Device Under Investigation (Total of Groups) | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/68 | 1/17 | 1/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 37/68 | 7/17 | 11/17 | 9/17 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Under Investigation (Total of Groups) (N=68) | Group 1 (N=17) | Group 2 (N=17) | Group 3 (N=17) | Group 4 (N=17)
spleen cyst (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
strangulated femoral hernia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Under Investigation (Total of Groups) (N=68) | Group 1 (N=17) | Group 2 (N=17) | Group 3 (N=17) | Group 4 (N=17)
ADE (Surgical and medical procedures) | 9 (12) | 4 (5) | 2 (2) | 1 (2) | 2 (3) — Adverse Device Effect
AE not device related (Surgical and medical procedures) | 28 (79) | 3 (13) | 9 (31) | 8 (11) | 8 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT06142578/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT06142578/ICF_001.pdf